CLINICAL TRIAL: NCT01250353
Title: The Use of Natural Latex Biomembrane in Ocular Surface Reconstruction and Pterygium
Brief Title: The Use of Natural Latex Biomembrane in Ocular Surface Reconstruction
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Erika Christina Canarim Martha de Pinho, RIbeirão Preto Faculty of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12416/05
Record Dates: First submitted 2010-11-24; First posted 2010-11-30 (Estimated); Last update posted 2010-11-30 (Estimated); Status verified 2009-12

CONDITIONS: Conjunctival Diseases; Pterygium
Keywords: ocular surface reconstruction; conjunctival healing; pterygium; latex biomembrane; pterygium surgery
MeSH Terms: conditions — Conjunctival Diseases; Pterygium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- conjunctival autograft (Experimental): The conjunctival autograft was performed after the pterygium surgery like usual technique.
  Interventions: Procedure: pterygium surgery
- latex biomembrane application (Experimental): The latex biomembrane was applied after pterygium surgery to recover the bare sclera area. This device was closed to conjunctiva with running suture anchored at some places to episclera. The sutures was removed at fourteenth day after surgery.
  Interventions: Procedure: pterygium surgery

INTERVENTIONS:
Procedure: pterygium surgery — pterygium was removed surgically
  Other Names: pterygium excision; prevention of pterygium recurrence

SUMMARY:
The main problem of ocular surface reconstruction is the lack of viable conjunctival tissue. The use of a biocompatible latex biomembrane in ocular surface healing, like post pterygium surgery, could be an alternative therapeutic resource to this process.

DETAILED DESCRIPTION:
The latex biomembrane is considered biocompatible and believed to promote neoformation of biological tissues. It also induces vascular neoformation and promotes extra cellular provisional matrix formation, fundamental steps for any kind of wound healing. In humans, it was successfully used in chronic cutaneous ulcer and otologic surgeries. In rabbits' eyes, the latex biomembrane was efficient in ocular surface reconstruction with adequate conjunctiva functional recovery, compared to bare sclera. To study the latex biomembrane action in human ocular surface, it was compared to conjunctival autograft in humans eyes. Considering the deficiency of adequate sized groups and the pterygium recurrences criteria differences, this study proposes the fibrovascular tissue growing measure like an auxiliary method of pos-operative evaluation. The biomembrane of natural latex seems to be efficient in ocular surface reconstruction and must be employed in future studies of other ocular pathologies. This material revealed to be a new source of therapeutic resort to external eye diseases and conjunctival replace in surgeries living bare sclera.

ELIGIBILITY:
Inclusion Criteria:

* symptomatic pterygium

Exclusion Criteria:

* any other ocular surface pathology, glaucoma, retinal disease, pregnancy, auto immune disease, severe systemic disease

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2006-06; Primary Completion 2007-06 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
change in fibrovascular tissue growing measure | twelve months
  The fibrovascular tissue growing measure was designed to be an auxiliary method of pos-operative evaluation. At the slit lamp, the pterygium or the fibrovascular growing tissue was measured related to anatomic limbus. To the scleral side was given negative value and to the cornea side was given positive value. The anatomic limbus was the zero in this scale. The results were compared at inicial stage and three, six and twelve months, to evaluate the progression and recurrence probability.

SECONDARY OUTCOMES:
pterygium recurrence | twelve months
  Pterygium recurrence was defined like fibrovascular tissue growing up to 1,5mm across the anatomic limbus.

CONTACTS AND LOCATIONS:
Overall Officials: Sidney JF Sousa, phD, Study Chair — Ribeirão Preto Faculty of Medicine
Locations (1):
- Erika Christina Canarim Martha de Pinho, Ribeirão Preto, São Paulo, Brazil

REFERENCES:
- [Background] Geggel HS, Friend J, Thoft RA. Conjunctival epithelial wound healing. Invest Ophthalmol Vis Sci. 1984 Jul;25(7):860-3. PMID 6735650
- [Background] PINHO, E.C.C.M. Uso de uma membrana derivada de látex natural na superfície ocular. Estudo experimental em coelhos. Dissertação. (Mestrado em Oftalmolgia). Ribeirão Preto, Universidade de São Paulo, 2003. p 96.
- [Background] PINHO, E.C.C.M.; FARIA E SOUSA, S.J.; CHAHUD, F.; LACHAT, J-J.; COUTINHO - NETTO, J. Uso experimental da biomembrana de látex na reconstrução conjuntival. Arquivos Brasileiros de Oftalmologia, v. 67, p. 27- 32, 2004.
- [Background] PINHO, E.C.C.M.; SEIXAS, G.C.O.; SOUZA-JUNIOR, E.N.; FARIA E SOUSA, S.J.; LACHAT, J-J.; COUTINHO - NETTO, J. The use of natural latex in human eye: technique description. In: Congresso Mundial de Oftalmologia, 2006a, São Paulo. Anais eletrônicos, código 2717.
- [Background] PINHO, E.C.C.M; FARIA E SOUSA, S.J.; SOUZA-JUNIOR, E.N.; SEIXAS, G.C.O.; LACHAT, J-J.; COUTINHO - NETTO, J. The use of natural latex in ocular surface, like tissue repair promoter, in pterygium excision. In: Congresso Mundial de Oftalmologia, 2006b, São Paulo. Anais eletrônicos, código 2150.